CLINICAL TRIAL: NCT06713928
Title: Effectiveness of Dog-Assisted Therapy on Compliance and Home Oral Hygiene Activities in Disabled Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jacopo Lanzetti, Dental Hygienist, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0000793
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Disabilities; Dog Therapy; Oral Hygiene, Oral Health
MeSH Terms: interventions — Oral Hygiene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hygiene with dog therapy (Experimental): use the DAT to support the oral hygiene procedures provided.
  Interventions: Other: Oral hygiene with dog therapy
- Oral hygiene without dog therapy (No Intervention): make oral hygiene without any type of support

INTERVENTIONS:
Other: Oral hygiene with dog therapy — The DAT session is divided into two phases: a pre-sitting phase in which the patient could interact with the dog, touching, caressing and playing with him, under the supervision of the dog-trainer. This phase lasted about 15 minutes. The second phase was a during-sitting phase in which the dog was in the chair, next to the patient, during the entire oral hygiene procedure, under the supervision of the dog-trainer.
  Arms: Oral hygiene with dog therapy

SUMMARY:
Recent scientific studies have shown how interaction with an animal can alleviate particular conditions of stress and conflict, thus representing a solid support for minor patients with social behavior problems or with physical or mental disabilities. In this co-therapy, a fundamental role is played by the relationship that is established between the human being and the animal, a very particular relationship capable of bringing about positive changes, in both members, but especially in the man who, benefiting from this push for change, can improve his own situation, whatever it is, and follow with greater interest and involvement the actual therapy activities proposed by the team that is following him.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to be between 5 and 16 years old;
* Patients with disability;
* Non-collaborating or with limited collaboration (Frankl Scale 1 or 2);
* Patients with a Plaque Control Record (PCR) of 40% or more;
* Patients with partial autonomy in home oral hygiene procedures.

Exclusion Criteria:

* Patients with fear of dogs;
* Patients with dog hair allergy;
* Patients with infectious disease;
* Tetraplegic and visually impaired subjects.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record (PCR) | 1 month
  PCR values the presence of dental plaque on the teeth

SECONDARY OUTCOMES:
Emotional record | 1 month
  the patient's perception was recorded using a graphic card that represents the moods of the moment of oral hygiene session

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided